CLINICAL TRIAL: NCT00286117
Title: An Open Randomised Clinical Study Comparing ARIMIDEX™ With NOLVADEX™ as Adjuvant Therapies in Post-Menopausal Women With Breast Cancer Already Being Treated With NOLVADEX for at Least Two Years
Brief Title: ITA - Clinical Study Comparing ARIMIDEX™ With NOLVADEX™ in Women With Breast Cancer Treated With NOLVADEX for at Least 2 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Francisco Sapunar, MD - Arimidex Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1033IT/0002; ITA
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

ARMS (2):
- 1 (Experimental): Anastrozole
  Interventions: Drug: Anastrozole
- 2 (Active Comparator): Tamoxifen
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — oral
  Other Names: Arimidex; ZD1033
  Arms: 1
Drug: Tamoxifen — oral
  Other Names: Nolvadex
  Arms: 2

SUMMARY:
The purpose of this study was to assess the difference in disease-free survival between post-menopausal women with hormone receptor-positive early breast cancer who switched from tamoxifen to anastrozole and those who continued on tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal status; age ≤75 years;
* histologically confirmed invasive breast cancer with metastases in the axillary lymph nodes;
* oestrogen receptor status positive or unknown;
* primary treatment (surgery +/- radiotherapy, +/- chemotherapy) completed

Exclusion Criteria:

* Clinical evidence of metastatic disease (including local or remote recurrence, even if the patient appeared to be in complete remission at the time of randomisation).

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 1998-03; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this analysis was to assess the difference in disease-free survival between post-menopausal women with hormone receptor-positive early breast cancer who switched from tamoxifen to anastrozole and those who continued on tamoxifen

SECONDARY OUTCOMES:
Assess the difference in overall survival/disease recurrence/safety and tolerability between post-menopausal women with hormone receptor-positive early breast cancer who switched from tamoxifen to anastrozole and those who continued to receive tamoxifen.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Arimidex Medical Science Director, MD, Study Director — AstraZeneca; Francesco Boccardo, MD, Principal Investigator — University and National Cancer Research Institute
Locations (25):
- Italy (25):
  - Research Site, Arezzo
  - Research Site, Bologna
  - Research Site, Casalpusterlengo
  - Research Site, Catania
  - Research Site, Chieti
  - Research Site, Ferrara
  - Research Site, Florence
  - Research Site, Forlì
  - Research Site, Genova
  - Research Site, Lugo
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Monserrato
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Pinerolo
  - Research Site, Roma
  - Research Site, Rovigo
  - Research Site, Sanremo
  - Research Site, Saronno
  - Research Site, Sassari
  - Research Site, Terni
  - Research Site, Torino
  - Research Site, Trieste
  - Research Site, Vicenza